CLINICAL TRIAL: NCT03479021
Title: Accuracy of Welch Allyn Spot™ Vision Screener to Detect Amblyogenic Factors in Developmentally Delayed Children
Brief Title: SPOT Vision Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital Colorado (Other)
Collaborators: Welch Allyn (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-1911 SPOT
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Vision Disorders
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: Welch-Allyn Spot Vision Screener — photograph of the eye

SUMMARY:
The purpose of this protocol is to determine if the Welch-Allyn Spot Vision Screener (SPOT) is effective at detecting various risk factors for poor vision in developmentally delayed children. These children have a higher percentage of vision disorders than the average population. The SPOT screen itself takes about six seconds to complete. It produces a photograph of the eye and a print out with amount of hyperopia, myopia, astigmatism and pupil size. The subject will have three SPOT screens around the time of their standard of care eye exam. The data obtained from the three SPOT screens will be compared among themselves for accuracy and to the findings of the clinical eye exam.

ELIGIBILITY:
Inclusion Criteria:

child over 4 months of age social, behavioral, physical, or other handicap unable to complete age-appropriate vision screening

Exclusion Criteria:

glaucoma post intraocular surgery microphthalmia other serious eye disorder inability to complete SPOT screener

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The children have various disabilities or delays to include: Attention Deficit Hyperactivity Disorder (ADHD), Autism Spectrum Disorder (ASD), chromosomal abnormalities such as Down Syndrome, Cerebral Palsy (CP), and mental retardation (MR).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
the SPOT will be effective in screening for amblyogenic risk factors | 12 months
  the Spot has a sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) necessary to appropriately perform visual triage in developmentally delayed children

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States